CLINICAL TRIAL: NCT00820131
Title: A Multicenter Prospective Randomized Trial on Chronic Pain After Inguinal Hernia Repair Using a Selfgrip-mesh
Brief Title: Chronic Pain After Inguinal Hernia Repair
Acronym: GRIP-ME
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Gerhard Prager, MD, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EK MUW 613/2007
Record Dates: First submitted 2009-01-08; First posted 2009-01-09 (Estimated); Last update posted 2014-12-09 (Estimated); Status verified 2009-01

CONDITIONS: Inguinal Hernia; Chronic Pain
MeSH Terms: conditions — Hernia, Inguinal; Chronic Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- 1 (Experimental)
  Interventions: Procedure: selfgrip mesh
- 2 (Active Comparator)
  Interventions: Procedure: lightweight mesh with suture fixation

INTERVENTIONS:
Procedure: selfgrip mesh — inguinal hernia repair using a selfgrip mesh
  Arms: 1
Procedure: lightweight mesh with suture fixation — inguinal hernia repair using a lightweight mesh with suture fixation
  Arms: 2

SUMMARY:
Chronic pain after inguinal hernia repair has become a major concern. Although tension-free Lichtenstein technique is used and new lightweight meshes have been developed, still up to 40 % of patients complain of some kind of pain even one year after surgery. The necessity of mesh-fixation using sutures, could be causative. However, current data do not provide evidence whether suture fixation in Lichtenstein repair might be the reason for chronic postoperative pain.

A newly developed selfgrip-mesh enables sutureless fixation of the mesh in open inguinal hernia repair. Hereby a polypropylene mesh is combined with a resorbable polylactic-acid gripping system. Thereby the rate of chronic postoperative pain could be decreased.

Two techniques of inguinal hernia repair will be evaluated:

1. open anterior mesh repair using conventional Lichtenstein technique (sutures for mesh-fixation)
2. open anterior mesh repair using a selfgrip mesh (polylactic-acid gripping system for mesh fixation)

Postoperative pain will be evaluated by visual analog scale and Mc Gill pain questionaire at the 10th day, as well as 3 and 15 months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* primary unilateral inguinal hernia
* 18 years and older

Exclusion Criteria:

* bilateral hernia
* recurrent hernia
* incarcerated hernia
* malignant disease within the last 5 years
* not able to understand the questionaire

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2008-01; Primary Completion 2013-01 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
chronic pain | 3 months, 15 months

SECONDARY OUTCOMES:
morbidity | 3 months, 15 months
recurrence rate | 3 months and 15 months
quality of life | 3 months and 15 months

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Prager, MD, Principal Investigator — Medical University of Vienna
Locations (7):
- Austria (7):
  - LKH Feldkirch, Dept. of Surgery, Feldkirch
  - Hospital Barmherzige Schwestern, Linz
  - LK Weinviertel Mistelbach, Surgical Department, Mistelbach
  - KH Göttlicher Heiland, Vienna
  - KFJ Hospital, Dept. of Surgery, Vienna
  - Medical University of Vienna, Dept. of Surgery, Vienna
  - KH Wiener Neustadt, Surgical Department, Wiener Neustadt